CLINICAL TRIAL: NCT02319525
Title: Individualized Patient Decision Making for Treatment Choices Among Minorities With Lupus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Jasvinder Singh, MD, MPH, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CE-1304-6631
Record Dates: First submitted 2014-11-05; First posted 2014-12-18 (Estimated); Results first posted 2017-01-31 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Systemic Lupus Erythematosus
Keywords: lupus nephritis; lupus; decision-making; minorities; immunosuppressive medications; decision-aid; treatment; Decision conflict; SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computerized patient decision-aid (Experimental): A computerized decision-aid showing benefits and harms of medications in words patients prefer
  Interventions: Other: Computerized patient decision-aid
- Usual care (lupus pamphlet) (Active Comparator): A handout/pamphlet from a non-profit organization on lupus and lupus medications (American College of Rheumatology [ACR])
  Interventions: Other: Usual care (lupus pamphlet)

INTERVENTIONS:
Other: Computerized patient decision-aid — The decision-aid contained information regarding lupus and lupus nephritis, its impact on patient lives and benefits and harms of lupus nephritis treatments, focused on immunosuppressive medications compared to each other. The content of the decision-aid allowed individualization based on patient preference for details on certain aspects, as well as the desire to view additional, optional sections of the decision-aid.
  Arms: Computerized patient decision-aid
Other: Usual care (lupus pamphlet) — Patient received the standard handout/pamphlet from a non-profit organization (American College of Rheumatology [ACR]) regarding lupus and its treatments, that explained risks and benefits of various treatments
  Arms: Usual care (lupus pamphlet)

SUMMARY:
The study will compare the efficacy of the usual education materials to individualized computerized decision guide on decision conflict of patients with lupus nephritis making treatment decisions regarding immunosuppressive therapies.

DETAILED DESCRIPTION:
The proposed study, a randomized controlled trial [RCT], will evaluate methods to assist minority lupus patients (African-Americans and Hispanics) to make shared decisions for the management of their lupus nephritis considering what is the best for them. We have developed an individualized patient decision guide that is culturally sensitive since it was developed solely based on the values, beliefs and preferences of minority patients. We will test the effectiveness of individualized decision aids in African-American and Hispanic lupus nephritis patients in a 2-arm randomized trial including 200 patients. We hypothesize that use of decision-aid will be associated with reduction in decisional conflict and more informed choice compared to usual care group (American College of Rheumatology [ACR] lupus pamphlet; co-primary effectiveness outcomes), both clinically meaningful and patient-centered outcomes. We chose the low-literacy decisional conflict scale as our primary outcome, since it is a validated measure, and the most commonly used outcome measure in decision aids RCTs. We use informed choice as a co-primary outcome, since this is conceptually most immediate to the intervention. It will measure whether in those with knowledge of risks and benefits of immunosuppressive drugs, patient values are concordant with their choice of immunosuppressive drug. Secondary outcomes include patient involvement in decision-making (concordance on control preference scale) and patient-physician communication (Interpersonal Processes of Care (IPC) score and analysis of audiotaped physician-patient Interaction (using the Active Patient Participation Coding Scheme (APPC)). Since we planned to recruit patients with current lupus nephritis flare (making current decision for an immunosuppressive drug) and with past lupus nephritis flares (making the same decision for a future lupus nephritis flare), two secondary outcomes (control preference scale for concordance of preferred and real role in deciding about immunosuppressive drugs and the audiotaped physician-patient interaction about immunosuppressive drugs) will be analyzed only in patients with current lupus nephritis flare, a subset of the entire cohort.

ELIGIBILITY:
Inclusion Criteria:

* adult female lupus nephritis patients, currently having a flare of lupus nephritis and considering change or initiation of an immunosuppressive medication (current flare) or had had flare of lupus nephritis in the past and at risk for a future lupus nephritis flare (future flare)

Exclusion Criteria:

* male; lupus but no lupus nephritis; change in lupus immunosuppressive treatment already made for current flare; end stage renal disease on dialysis; renal transplant or candidate for a renal transplant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jasvinder Singh, MBBS, MPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh JA, Fraenkel L, Green C, Alarcon GS, Barton JL, Saag KG, Hanrahan LM, Raymond SC, Kimberly RP, Leong AL, Reyes E, Street RL Jr, Suarez-Almazor ME, Eakin GS, Marrow L, Morgan CJ, Caro B, Sloan JA, Jandali B, Garcia SR, Grossman J, Winthrop KL, Trupin L, Dall'Era M, Meara A, Rizvi T, Chatham WW, Yazdany J. Individualized decision aid for diverse women with lupus nephritis (IDEA-WON): A randomized controlled trial. PLoS Med. 2019 May 8;16(5):e1002800. doi: 10.1371/journal.pmed.1002800. eCollection 2019 May. PMID 31067237
- [Derived] Singh JA, Shah N, Green C. Individualized patient decision-aid for immunosuppressive drugs in women with lupus nephritis: study protocol of a randomized, controlled trial. BMC Musculoskelet Disord. 2017 Jan 31;18(1):53. doi: 10.1186/s12891-017-1408-5. PMID 28143529

RESULTS

PARTICIPANT FLOW:
Groups:
- Decision Aid: Participants received decision aid tool providing information about medication choices for lupus nephritis
- Pamphlet: Participants received the standard American College of Rheumatology lupus pamphlet
Period: Overall Study
Arm/Group | Decision Aid | Pamphlet
Started | 153 | 148
Primary Research Completion | 151 | 147
Completed | 151 | 147
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Decision Aid | Pamphlet | Total
Number analyzed (Participants) | 151 | 147 | 298
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 148 | 146 | 294
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Full Range); unit: Years] | 37.1 [19 to 69] | 37.6 [19 to 66] | 37.3 [19 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 147 | 298
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Not answered | 2 | 0 | 2
  Asian | 11 | 9 | 20
  Hispanic/Latino | 41 | 37 | 78
  Non-Hispanic Black | 70 | 71 | 141
  Non-Hispanic White | 20 | 24 | 44
  Other | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 151 | 147 | 298
Decisional conflict [Mean (Standard Deviation); unit: units on a scale] — The Decisional Conflict Scale is a patient self-administered, validated measure of decisional conflict, a state of uncertainty about a course of action. Scores range from 0 (no decisional conflict) to 100 (extremely high decisional conflict).
  units on a scale | 33.37 (29.55) | 37.48 (29.85) | 35.4 (29.72)
Knowledge about immunosuppressives [Number; unit: participants] — Patients were asked 20 true/false questions regarding lupus nephritis and immunosuppressive drugs. Patients answering at least 75% of questions correctly were considered to have "adequate" knowledge about immunosuppressives. Those answering fewer than 75% of questions correctly were considered to have "inadequate" knowledge.
  participants
    Adequate Knowledge | 90 | 89 | 179
    Inadequate Knowledge | 61 | 58 | 119

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Decisional Conflict Scale Scores
Description: Patient self-administered, validated measure of decisional conflict, most commonly used as the primary outcome in RCTs of decision aids (change score). The score ranges from 0 (no decisional conflict) to 100 (extreme decisional conflict). Decisional conflict represents a state of uncertainty about a choice or course of action and is more likely in situations involving high-stakes choices with important potential gains and losses, value tradeoffs in selecting a choice or a course of action (vs. the alternative) or uncertain outcomes.
Time Frame: Baseline and after viewing the decision-aid or the standard hand-out (pamphlet) on the same visit as the intervention (preferred) but before treatment decision-making (usually within 1 week)
Population: All participants who received either the Decision Aid or Pamphlet
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Decision Aid | Pamphlet
Number analyzed (Participants) | 151 | 147
units on a scale | 21.80 (30.89) | 12.69 (24.41)
Statistical Analysis 1: Comparison: Decision Aid vs Pamphlet; Test type: Superiority or Other; p = 0.005, t-test, 2 sided

2. Primary Outcome: Informed Choice (Validated Instruments for Values Regarding Immunosuppressives, Knowledge About Immunosuppressives, and Treatment Decision-making)
Description: Concordance between values related (for or against starting) immunosuppressive drugs with patients' decision (to start or not start) immunosuppressive drugs, in those with adequate knowledge about benefits/harms of immunosuppressive drugs, assessed using validated instruments for values regarding immunosuppressive drugs, knowledge about immunosuppressive drugs, and treatment decision-making (patient's decision to start immunosuppressive drug).
Time Frame: After viewing the guide or standard hand-out on the same visit as the intervention (preferred) but before treatment decision-making (usually within 1 week)
Population: All participants who received either the Decision Aid or Pamphlet.
Measure: Number; unit: participants
Arm/Group | Decision Aid | Pamphlet
Number analyzed (Participants) | 151 | 147
participants
  Informed Choice Made | 62 | 46
  No Informed Choice | 89 | 101
Statistical Analysis 1: Comparison: Decision Aid vs Pamphlet; Test type: Superiority or Other; p = 0.08, Chi-squared — We compared informed choice vs. no informed choice made between the decision aid and the pamphlet groups

3. Secondary Outcome: Control Preferences Scale: Patient Participation in Decision-making
Description: This scale assessed how much decision-making control they would like to have versus actually experienced. There are 5 responses for 5 control options: active, active shared, collaborative, passive shared and passive, which were collapsed into active (active, active shared), collaborative, and passive (passive shared and passive), as previously (and pre-specified). Concordance was assessed between desired and actual role played by each patient. We present these data for patients with current flare only, since only they were making a decision about the immunosuppressive drugs; patients with past lupus flare were not included in the denominator.
Time Frame: as for outcome 2
Population: Only participants having a current lupus nephritis and requiring immunosuppressive medication change/initiation or participants with newly diagnosed lupus nephritis starting an immunosuppressive medication.
Measure: Number; unit: participants
Arm/Group | Decision Aid | Pamphlet
Number analyzed (Participants) | 35 | 33
participants
  Concordance between roles | 33 | 28
  No concordance between roles | 2 | 5
Statistical Analysis 1: Comparison: Decision Aid vs Pamphlet; We compared concordance between preferred and actual roles vs. no concordance between roles between decision aid and pamphlet; Test type: Superiority or Other; p = 0.252, Chi-squared

4. Secondary Outcome: Patient Physician Communication (Interpersonal Processes of Care (IPC)
Description: This was assessed using the interpersonal processes of care (IPC), an 18-item validated patient-reported measure of patient-physician communication and care processes. The score ranges from 18 (worst) to 90 (best) and the scale is a patient-reported measure of patient-physician communication and care processes.
Time Frame: After viewing the guide or standard hand-out on the same visit as the intervention (preferred) (usually within 1 week)
Population: All participants who received either the Decision Aid or Pamphlet.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Decision Aid | Pamphlet
Number analyzed (Participants) | 149 | 147
units on a scale | 83.64 (7.69) | 83.06 (7.28)
Statistical Analysis 1: Comparison: Decision Aid vs Pamphlet; Test type: Superiority or Other; p = 0.504, t-test, 2 sided

5. Secondary Outcome: Analysis of Audiotaped Physician-patient Interaction (Using the Active Patient Participation Coding Scheme (APPC)): Doctor Patient-centered Communication
Description: This was done by analyzing the audio-recorded patient-physician discussion in patients with current lupus nephritis flare. The APCC is a validated instrument to measure 'active patient participation.' APCC assesses indicators and facilitators of patient participation. The unit of coding is the utterance, the oral analogue of a sentence. The range is 0 to unlimited. Patient participation is measured by the number of questions, number of concerns expressed, and act of assertiveness (e.g., preferences, introducing topics, making requests). These are 'active' forms of participation because of their influence on clinician behavior and the structure and content of the consultation. The APPC also assess clinician behaviors that facilitate and support patient participation, partnership-building and supportive talk (e.g., reassurance, empathy). We present doctor patient-centered communication. higher scores indicates better patient participation and communication.
Time Frame: After viewing the guide or standard hand-out on the same visit as the intervention (preferred) (usually within 1 week)
Population: Only participants having a current lupus nephritis and requiring immunosuppressive medication change/initiation or participants with newly diagnosed lupus nephritis starting an immunosuppressive medication, who also agreed for an audio-recorded conversation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Decision Aid | Pamphlet
Number analyzed (Participants) | 16 | 17
units on a scale | 5.1 (2.1) | 3.7 (1.9)
Statistical Analysis 1: Comparison: Decision Aid vs Pamphlet; Test type: Superiority or Other; p = 0.06, t-test, 2 sided

6. Secondary Outcome: Acceptability (Number of Participants Rating Each Statement as "Excellent")
Description: Acceptability of the decision-aid (information quality and quantity, presentation style and usefulness) was assessed using a validated acceptability survey on 4-point scale ranging from "excellent" to "poor" (response options were: excellent, good, fair and poor). The number of patients rating each of the five statements as "excellent" (vs. other ratings) was compared between the two treatment arms.
Time Frame: After viewing the guide or standard hand-out on the same visit as the intervention (preferred) (usually within 1 week)
Measure: Count of Participants; unit: Participants
Arm/Group | Decision Aid | Pamphlet
Number analyzed (Participants) | 151 | 147
Participants
  Impact of lupus nephritis | 74 | 49
  Risk factors | 64 | 40
  Medication options | 76 | 49
  Evidence about medications | 71 | 35
  Studies about other patients | 64 | 32
Statistical Analysis 1: Comparison: Decision Aid vs Pamphlet; statistical analysis comparing the decision-aid vs. pamphlet for patient rating of acceptability of information and presentation related to the "Impact of lupus nephritis"; Test type: Superiority or Other; p = 0.006, Chi-squared
Statistical Analysis 2: Comparison: Decision Aid vs Pamphlet; statistical analysis comparing the decision-aid vs. pamphlet for patient rating of acceptability of information and presentation related to the "Risk factors"; Test type: Superiority or Other; p = 0.006, Chi-squared
Statistical Analysis 3: Comparison: Decision Aid vs Pamphlet; statistical analysis comparing the decision-aid vs. pamphlet for patient rating of acceptability of information and presentation related to the "medication options"; Test type: Superiority or Other; p = 0.003, Chi-squared
Statistical Analysis 4: Comparison: Decision Aid vs Pamphlet; statistical analysis comparing the decision-aid vs. pamphlet for patient rating of acceptability of information and presentation related to the "evidence about medications"; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 5: Comparison: Decision Aid vs Pamphlet; statistical analysis comparing the decision-aid vs. pamphlet for patient rating of acceptability of information and presentation related to the "study about other patients"; Test type: Superiority or Other; p < 0.001, Chi-squared

7. Secondary Outcome: Feasibility (Number of Participants Rating the Feasibility of Using Decision-aid or Pamphlet- Referred to as Education Guide in This Statement)
Description: Feasibility of the decision-aid vs. pamphlet was assessed using a single statement "The education guide was easy to use". Patients rated this on 5-point ordinal scale ranging from "strongly agree" to "strongly disagree" (response options were: strongly agree, agree, neither agree nor disagree, disagree, strongly disagree). The number of patients was compared between the two treatment arms.
Time Frame: After viewing the guide or standard hand-out on the same visit as the intervention (preferred) (usually within 1 week)
Population: One patient from pamphlet group did not respond to this question, therefore valid responses from pamphlet were 146, not 147
Measure: Count of Participants; unit: Participants
Arm/Group | Decision Aid | Pamphlet
Number analyzed (Participants) | 151 | 146
Participants
  Strongly Disagree | 1 | 3
  Disagree | 1 | 13
  Neither Agree nor Disagree | 73 | 74
  Agree | 75 | 55
  Strongly Agree | 1 | 1
  Missing | 0 | 1
Statistical Analysis 1: Comparison: Decision Aid vs Pamphlet; The test of significance compared all the rows, i.e., all response options for the statement; Test type: Superiority or Other; p = 0.006, Chi-squared

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Decision Aid | Pamphlet
All-Cause Mortality (participants affected / at risk) | 1/151 | 1/147
Serious Adverse Events (participants affected / at risk) | 1/151 | 1/147
Other Adverse Events (participants affected / at risk) | 0/151 | 0/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decision Aid (N=151) | Pamphlet (N=147)
Right ventricular failure (Vascular disorders) | 1 (1) | 0 (0) — 1. Decision-aid: Patient with mitral regurgitation died due of right ventricular failure after cardiovascular surgery (Day 53).
Subarachnoid hemorrhage (Vascular disorders) | 0 (0) | 1 (1) — 1. Pamphlet: Subarachnoid hemorrhage from posterior circulation aneurysm. Patient died due to central herniation (Day 22)

LIMITATIONS AND CAVEATS:
1. Study findings may not be generalizable to men with lupus, since we studied only women
2. It remains to be seen whether our decision-aid can be used by lupus patients with non-renal manifestations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No